CLINICAL TRIAL: NCT00003436
Title: Medical Research Council Working Party on Leukaemia in Childhood Acute Myeloid Leukaemia Trial 12
Brief Title: Combination Chemotherapy With or Without Bone Marrow Transplantation in Treating Children With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066463; MRC-LEUK-AML12CH; EU-98010
Record Dates: First submitted 1999-11-01; First posted 2003-04-30 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2000-12

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: untreated childhood acute myeloid leukemia and other myeloid malignancies; childhood acute promyelocytic leukemia (M3); refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; secondary myelodysplastic syndromes; childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Anemia, Refractory, with Excess of Blasts | interventions — Amsacrine; Asparaginase; Cytarabine; Daunorubicin; Etoposide; Methotrexate; Mitoxantrone; Hydrocortisone

INTERVENTIONS:
Drug: amsacrine
Drug: asparaginase
Drug: cytarabine
Drug: daunorubicin hydrochloride
Drug: etoposide
Drug: methotrexate
Drug: mitoxantrone hydrochloride
Drug: therapeutic hydrocortisone
Procedure: allogeneic bone marrow transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with bone marrow transplantation may allow doctors to give higher doses of chemotherapy and kill more cancer cells. It is not yet known whether chemotherapy is more effective with or without bone marrow transplantation for acute myeloid leukemia.

PURPOSE: Randomized phase III trial to compare the effectiveness of chemotherapy with or without bone marrow transplantation in treating children who have acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare two induction schedules with respect to achievement and duration of remission, survival, toxicity, and supportive care requirements in children with previously untreated acute myeloid leukemia.
* Compare 4 versus 5 courses of treatment in total (where the final course is either chemotherapy or bone marrow transplantation) with respect to remission duration, relapse rates, deaths in remission, and overall survival in these patients.
* Compare the value of allogeneic bone marrow transplantation versus conventional chemotherapy with respect to remission duration, relapse rates, deaths in remission, and overall survival in these patients.
* Reduce toxicity without compromising survival by restricting the number of patients receiving bone marrow transplant in this study.

OUTLINE: This is a randomized study. Patients are first randomized to one of two induction treatment arms.

* Induction Arm I: Patients receive 2 courses of cytarabine IV push every 12 hours on days 1-10 or 1-8 (20 or 16 doses); daunorubicin IV over 6 hours on days 1, 3, and 5; and etoposide IV over 4 hours on days 1-5 (5 doses).
* Induction Arm II: Patients receive 2 courses of mitoxantrone IV over 6 hours on days 1, 3, and 5; cytarabine IV push every 12 hours on days 1-10 or 1-8 (20 or 16 doses); and etoposide IV over 4 hours on days 1-5 (5 doses).

Patients with no CNS disease at diagnosis receive 3 courses of triple intrathecal therapy (methotrexate, cytarabine, and hydrocortisone), one after each of the first 3 courses of chemotherapy. Patients with CNS disease receive at least 6 courses of intrathecal therapy (2 courses per week), then monthly courses until the final course of chemotherapy is complete.

Patients in complete response after induction course 2 continue on this study. Patients not in complete response after induction course 2 are taken off study and are eligible for the current Medical Research Council (MRC) refractory/relapse study or another therapy.

Course 3: All patients continuing on this study receive amsacrine IV over 1 hour daily on days 1-5, cytarabine continuous IV infusion daily on days 1-5, and etoposide IV over 4 hours on days 1-5 as course 3. After course 3, patients are assigned to two risk groups: good risk patients, and standard and poor risk patients.

Standard and poor risk patients with no matched sibling donor and good risk patients are then further randomized to consolidation in arms I or II.

* Arm I: Patients receive mitoxantrone IV over 6 hours on days 1-5 and cytarabine IV over 2 hours every 12 hours on days 1-3 (4 courses of chemotherapy total).
* Arm II: Patients receive cytarabine IV over 3 hours every 12 hours on days 1, 2, 8, and 9, and asparaginase subcutaneous infusion 3 hours after completion of the last cytarabine doses on days 2 and 9, followed by a course of mitoxantrone and cytarabine as in arm I (5 courses of chemotherapy total).

Standard and poor risk children with matched sibling donor are randomized to arms III or IV.

* Arm III: Patients receive no consolidation treatment (3 courses of chemotherapy total) plus bone marrow transplantation.
* Arm IV: Patients receive cytarabine and asparaginase as in arm II (4 courses of chemotherapy total) plus bone marrow transplantation.

Patients are followed for at least 1 year.

PROJECTED ACCRUAL: Approximately 2,000 patients will be accrued into this study over 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* One of the following diagnoses:

  * Histologically confirmed de novo or secondary acute myeloid leukemia (AML)
  * Aggressive myelodysplastic syndromes (refractory anemia with excess blasts (RAEB) and RAEB in transformation) for which intensive AML therapy is considered appropriate
  * Acute promyelocytic leukemia (should also be entered into protocol MRC-ATRA)
* No chronic myeloid leukemia in blast transformation
* Must be considered suitable for intensive chemotherapy

PATIENT CHARACTERISTICS:

Age:

* Under 16

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No other concurrent active malignancy

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy for leukemia

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2000 (Estimated)
Dates: Start 1998-07; Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim O.B. Eden, MB, BS, FRCPE, FRCP, FRCPCH, F, Study Chair — The Christie NHS Foundation Trust
Locations (1):
- Christie Hospital N.H.S. Trust, Manchester, England, United Kingdom

REFERENCES:
- [Background] Gibson BE, Wheatley K, Hann IM, Stevens RF, Webb D, Hills RK, De Graaf SS, Harrison CJ. Treatment strategy and long-term results in paediatric patients treated in consecutive UK AML trials. Leukemia. 2005 Dec;19(12):2130-8. doi: 10.1038/sj.leu.2403924. PMID 16304572
- [Background] Burnett AK, Hills RK, Goldstone AH, et al.: The impact of transplant in AML in 2nd CR: a prospective study of 741 in the MRC AML 10 and 12 trials. [Abstract] Blood 104 (11): A-620, 2004.